CLINICAL TRIAL: NCT01874587
Title: Phase III Trial Testing the Benefit of Intensity-modulated Radiotherapy With Weekly Replanifications Versus Intensity Modulated Radiotherapy With Only One Planification in Locally Advanced Oropharynx Carcinoma for Decreasing Xerostomia
Brief Title: Adaptative Radiotherapy to Decrease Xerostomia in Oropharynx Carcinoma
Acronym: ARTIX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-RdC-ORL-Th; 2012-A00426-37 (Registry Identifier: ANSM)
Record Dates: First submitted 2013-04-25; First posted 2013-06-11 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Oropharynx Cancer
Keywords: Adaptative radiotherapy; oropharynx carcinoma; xerostomia
MeSH Terms: conditions — Oropharyngeal Neoplasms; Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard radiotherapy (No Intervention): single pre-treatment planning before radiotherapy
- adaptative radiotherapy (Experimental): adaptive Radiotherapy based on a weekly replanning
  Interventions: Radiation: adaptative radiotherapy

INTERVENTIONS:
Radiation: adaptative radiotherapy — weekly replanning
  Arms: adaptative radiotherapy

SUMMARY:
The Phase III study will include 174 patients with locally advanced oropharynx carcinoma, receiving all arc-IMRT (Intensity-Modulated Radiation Therapy) (70 Gy) with concomitant systemic therapy. Two arc-IMRT treatment arms will be compared: one "standard" arm based on the use of a single pre-treatment planning and one "experimental" arm (adaptive RT) based on a weekly replanning to spare the salivary glands. The main objective is to increase by 25% the salivary flow (Parafilm) 12 months after RT thanks to adaptive RT, while not decreasing local control. The secondary objectives are to increase the salivary flow (scintigraphy), reduce xerostomia, acute and late toxicities (Eisbruch questionnaire, MDAS-HN, v.4 CTCAE), while maintaining local control (stopping rule of the trial if difference>15%). 174 patients will be included in 6 French centers for 2 years and followed for 2 years. The HPV (Human Papillomavirus) status will be identified and the tumors frozen. A central IMRT QA (Quality Assurance) will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced non-metastatic carcinoma of the oropharynx limited to T3 and T4 (whatever the N) and N2-N3 (whatever the T)(AJCC stage III-IV)
2. Age ≥ 18 years and ≤ 75 years
3. Performance status (WHO ≤ 2)
4. Renal, hepatic and cardiovascular functions allowing systemic treatment administration
5. Adapted stomatologic care
6. Signed informed consent form
7. Membership or beneficiary of a national insurance scheme

Exclusion Criteria:

1. Both parotids totally included in the target volume
2. Stages T1 or T2 with positive node disease N1
3. Neoadjuvant chemotherapy
4. Exereses of primitive tumor and/or nodes
5. History of other cancer within 5 years (except for basocellular epithelioma and cervical)
6. Previous neck radiotherapy
7. Platinum salts, 5FluoroUracile (5FU) agents or cetuximab chemotherapy considerations
8. Unstable diseases (cardiovascular, renal, pulmonary, systemic lupus or sclerodermia)incompatible with study participation
9. Patient participating in other therapeutic trial with experimental drug, 30 days before the inclusion.
10. Patient already recruited in another biomedical research ( non interventional study is authorized)
11. Pregnant or breast feeding patients
12. Patient deprived of liberty, under tutorship, guardianship or placed under judicial protection
13. Patient is deemed incapable of giving informed consent
14. Patients who, for family, social, geographic or psychological reasons, cannot be adequately followed up and/or are incapable of undergoing regular controls.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Salivary flow measure | 12 months after the end of radiotherapy
  The salivary flow is measured after stimulation with Parafilm at the time of inclusion and then 12 months after the end of radiotherapy.

SECONDARY OUTCOMES:
Xerostomia | From before treatment to 24 months after the end of radiotherapy
  salivary flow measured after stimulation before treatment, 6months, 18 months and 24 months after the end of radiotherapy Eisbruch's questionnaire before treatment, at 3, 6, 12, 18 and 24 months after the end of radiotherapy
Salivary flow | Before treatment and 12 months after the end of radiotherapy
  measured by scintigraphy
Local control | 2 years
  analysed according stages T and N, HPV status
Early and late toxicities | From beginning of the radiotherapy up to 2 years after the end of radiotherapy
  early toxicity : weekly assessment during radiotherapy until 3 months after the end late toxicity : 6, 12, 18 and 24 months after the end of radiotherapy
Survival | 2 years
  overall and disease free survival
Head and Neck functionality | Before treatment to 24 months after the end of radiotherapy
  MDASI-HN questionnaire before treatment, 3, 6, 12, 18 and 24 months after the end of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Renaud De Crevoisier, MD, Principal Investigator — Centre Eugène Marquis - Rennes - France
Locations (11):
- France (11):
  - Clinique Claude Bernard, Albi
  - Clinique Pasteur - Saint Esprit, Brest
  - CRLCC Baclesse, Caen
  - CRLCC Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CRLCC Antoine Lacassagne, Nice
  - CHU de la Milétrie, Poitiers
  - Centre Eugene Marquis, Rennes
  - CRLCC Henri Becquerel, Rouen
  - Centre Paul Strauss, Strasbourg
  - CHU Tours, Tours

REFERENCES:
- [Derived] Castelli J, Thariat J, Benezery K, Hasbini A, Gery B, Berger A, Liem X, Guihard S, Chapet S, Thureau S, Auberdiac P, Pommier P, Ruffier A, Perrier L, Devillers A, Campillo-Gimenez B, de Crevoisier R. Weekly Adaptive Radiotherapy vs Standard Intensity-Modulated Radiotherapy for Improving Salivary Function in Patients With Head and Neck Cancer: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2023 Aug 1;9(8):1056-1064. doi: 10.1001/jamaoncol.2023.1352. PMID 37261806